CLINICAL TRIAL: NCT05010915
Title: Theta Burst Stimulation, Transcranial Magnetic Stimulation, Late Life Depression, Suicidal Ideation, Functional Magnetic Resonance Imaging, Dorsolateral Prefrontal Cortex, Ventrolateral Prefrontal Cortex
Brief Title: TBS,TMS, Suicidal Ideation, Magnetic Resonance Imaging, Dorsolateral Prefrontal Cortex, Ventrolateral Prefrontal Cortex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202002467A3
Record Dates: First submitted 2021-07-02; First posted 2021-08-18 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2023-08

CONDITIONS: Late Life Depression
Keywords: TMS; TBS
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dorsolateral prefrontal cortex (Experimental): 1. Age > 50 years.
  2. Major depressive disorder (MDD).
  3. Right handiness
  4. with a score ≥ 12 on the Beck Scale of Suicidal Ideation (BSSI) and a score of at least 3 on Question #3 (Suicide: 3 ideas and gestures of suicide) of the HAMD
  Interventions: Device: Transcranial magnetic stimulation
- ventrolateral prefrontal cortex (Experimental): 1. Age > 50 years.
  2. Major depressive disorder (MDD).
  3. Right handiness
  4. with a score ≥ 12 on the Beck Scale of Suicidal Ideation (BSSI) and a score of at least 3 on Question #3 (Suicide: 3 ideas and gestures of suicide) of the HAMD
  Interventions: Device: Transcranial magnetic stimulation
- sham comparator (Placebo Comparator): 1. Age > 50 years.
  2. Major depressive disorder (MDD).
  3. Right handiness
  4. with a score ≥ 12 on the Beck Scale of Suicidal Ideation (BSSI) and a score of at least 3 on Question #3 (Suicide: 3 ideas and gestures of suicide) of the HAMD
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial magnetic stimulation

SUMMARY:
Transcranial magnetic stimulation (TMS) is a noninvasive brain stimulation technique, its approved therapeutic indication is high-frequency stimulation to the left dorsolateral prefrontal cortex (DLPFC) for treatment resistant.

DETAILED DESCRIPTION:
investigators design a prospective three-year study to exam the effect of TBS on reducing suicidality targeted at left DLPFC vs VLPFC, and guided by task fMRI neuronavigation and sham. Investigators will adopt personalized left DLPFC and VLPFC localization from baseline task fMRI data. Due to the global brain atrophic changes in the older adults, this issue has been even more important. Investigators will enroll 163 late life depression cases, they will be randomly allocated to either DLPFC group (65 cases), or VLPFC group (65 cases) and sham group (33 cases). To sum up, investigators seek to evaluate the impact of an acute course of TBS guided by tsked fMRI neuronavigation on suicidal ideation, and through follow-up for 6 months, investigators expect to examine (1) suicidal ideation, structural and functional brain differences, inflammatory markers pre/post TBS treatment, explore the link between the mechanism underlying of TBS on brain connectivity and therapeutic effects (2) Association of suicide ideation and neurocognitive function, inflammatory factors and brain imaging data. Exploratory analysis will assess suicide ideation as mediator in the association of neurocognitive deficit and functional connectivity or neurocognitive deficit as mediator in the association of suicide ideation and brain imaging data (3) The trajectories of suicidal ideation in late life depression, to analysis whether the association of cognitive dysfunction and suicidal ideation occurs across time and the prediction of neurocognitive function.(4) Explore the association of suicidal ideation the depression severity, to test if suicidal ideation could be an independent treatment target (5) Investigate the plausible predictors of neuropsychological profiles or neuroimaging findings associated to the effect of TBS in reducing suicidal ideation, which could provide a more efficient strategy for suicide prevention in the elder.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years.
2. Major depressive disorder (MDD).
3. Right handiness
4. with a score ≥ 12 on the Beck Scale of Suicidal Ideation (BSSI) and a score of at least 3 on Question #3 (Suicide: 3 ideas and gestures of suicide) of the HAMD

Exclusion Criteria:

1. Inability to provide informed consent.
2. Dementia, as defined by MoCA 23/24. Other major mental or current psychotic symptoms
3. Active current suicidal intent as evidenced or the endorsement of an actual attempt, interrupted attempt,
4. Have known preexisting noise-induced hearing loss, concurrent treatment with ototoxic medications, or with cochlear implants are on medications known to lower seizure threshold.
5. Alcohol or other substances abuse of or dependence on within the past 3 months Organic brain, head trauma,
6. Elevated risk of seizure due to TBI
7. Participation in concurrent clinical trial
8. Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
9. Unstable medical illness, including delirium, malignancy, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management. Unstable cardiac disease or recent (<3m) myocardial infarction
10. Mental implement in the brain, claustrophobia
11. Ever received ECT, TMS Consent procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 125 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Beck Scale for Suicide Ideation (BSSI) at baseline | baseline(1 week before treatment)
  the severity of suicide ideation(the score range from 0-38,the higher score indicates higher severity.
Beck Scale for Suicide Ideation (BSSI)at the 1st month | the 1st month (4 weeks after baseline)
  the severity of suicide ideation(the score range from 0-38,the higher score indicates higher severity)
Beck Scale for Suicide Ideation (BSSI)at the 3rd month | the 3rd month(12 weeks after baseline)
  the severity of suicide ideation(the score range from 0-38,the higher score indicates higher severity)
Beck Scale for Suicide Ideation (BSSI)at the 6th month | the 6th month(24 weeks after baseline)
  the severity of suicide ideation(the score range from 0-38,the higher score indicates higher severity)

SECONDARY OUTCOMES:
Geriatric Depression Scale | baseline(1 week before treatment), the 1st month(4 weeks after baseline), the 3rd moth(12 weeks after baseline), and the 6th month(24 weeks after baseline)
  the severity of depression(the score range from 0-15,the higher score means worse outcome)
structural and functional connectivity | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  Brain MRI connectivity change
MRI T1 | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  Brain structural volumes (cm)
functional MRI (resting-state/biological motion task) - BOLD signal | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  Blood-oxygen-level-dependent (BOLD) signal is a measurement used in fMRI which reflects the neural activity.
Diffusion Tensor Imaging (DTI) - FA | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  Fractional anisotropy (FA) is a measurement used in DTI, which reflects the movement of water molecules. FA ranges from 0 to 1, the higher FA value may represent more intact axons.reflects the neural activity.
Verbal Learning & Memory: | baseline(1 week before treatment), the 1st month(4 weeks after baseline) and the 6th month(24 weeks after baseline)
  Word list of Wechsler Memory Scale-III Face memory task
Interleukin-1 | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  IL-1
Interleukin-2 | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  IL-2
Interleukin-6 | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  IL-6
Interleukin-10 | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  IL-10
Tumor necrosis factor | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  TNF-α
Interleukin-1β | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  IL-1β
C-Reactive protein | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  CRP
cortisol | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  cortisol
thyrotropin | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  TSH
Brain-derived neurotrophic factor | baseline(1 week before treatment), the 1st month(4 weeks after baseline)
  BDNF

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Hua Lee, Study Chair — ChungGung memorial hospital
Locations (1):
- "MAGSTIM" Repetitive transcranial magnetic stimulator(rTMS) System, Taoyuan District, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: No